CLINICAL TRIAL: NCT04862169
Title: Strengthening Palliative Care in Primary Health Care Through Knowledge Enhancement (SPARK) for Nurses in Yogyakarta: A Randomized Control Trial
Brief Title: Strengthening Palliative Care in Primary Health Care Through Knowledge Enhancement
Acronym: SPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Martina Sinta Kristanti, Principle Investigator, Assistant Professor, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPARK project 2021
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Palliative Care; Nurse; Community Health Services
Keywords: Palliative care; Nurses; Indonesia; Primary Health Center; SPARK Indonesia

STUDY DESIGN:
Intervention Model Description: The intervention on this RCT is SPARK (Sinau PAlliative Rame-rame bareng eLOK) OR Strengthening PAlliative caRe in the community by enhancing nurses' Knowledge). This is an educational intervention using an online method with learning method system (LMS) eLOK hosted by Universitas Gadjah Mada Yogyakarta (Affiliation of authors' team). The intervention includes online discussions and access to eLOK for study materials (modules and videos).
Who Masked: Participant, Investigator
Masking Description: Allocation concealment will use sealed envelopes. Randomization will be done by concealing a piece of paper that has the phrase "Intervention (SPARK)" or "Control (MODULE only)" which will be placed inside a thick envelope. The outside of the envelopes will be labelled with the sequence number. After a participant has been enrolled into the study and consented, the next sequence numbered envelope on the stack will be opened to determine the study group that the subject will enter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): In the control group, they will only receive electronic version of the modules. They are able to access the module on their own devices.
  The observation arm will receive the link of eLOK at the end of data collection and follow-ups (week 14). With this link, then they are able to access modules, videos and case studies provide in SPARK.
  Interventions: Other: electronic version of the modules
- Intervention group (Experimental): The intervention on this RCT is an educational training program: SPARK (Strengthening PAlliative caRe in the community by enhancing nurses' Knowledge). This is an educational intervention using an online method with learning method system (LMS) eLOK hosted by Universitas Gadjah Mada Yogyakarta (Affiliation of authors' team). The intervention includes online discussions and access to eLOK for study materials (modules and videos) and some synchronous meetings.
  Interventions: Other: educational intervention (SPARK)

INTERVENTIONS:
Other: educational intervention (SPARK) — There are 3 modules with 11 chapters. These topics were considered as the most relevant topics for implementation of palliative care for PHC nurses. Also, topics were selected based on our previous literature review of the previous study on the content of PHC nurses training program.
  The first module is the introduction. This consists of three chapters: introduction, support system and effective communication. Total reading time is estimated to be one hour. The second module is about the nursing approach in palliative care. It is estimated to be completed in around 2 hours and 15 minutes. The last module is about end of life care.
  The participants are expected to access this module before the scheduled synchronous mode. Modules will be provided in the electronic version, so that participants are able to download and read them on their own devices. We are also providing video as trigger for case study discussion
  Arms: Intervention group
Other: electronic version of the modules — electronic version of the modules
  Arms: Control group

SUMMARY:
The implementation of palliative care has been started in Indonesia since 2007. This was declared by Ministry of health regulation (SK Menkes no 812/Menkes/SK/2007). However, there has been a slow development in palliative care compared to other Asian countries. One of the reasons is the lack of knowledge and skills among health care professionals in Indonesia.

Primary Heath Center (PHC) is at the frontline in the health care system in Indonesia to provide care for patients. Its function is especially important in the Universal Health Coverage era. Studies have shown that PHC's nurses' knowledge on palliative care is still limited since the integration of palliative care into the nursing curriculum just started 2-3 years ago. Also, this curriculum integration is still limited in some Universities. Continuing nursing education (CNE) is one of the ways to enhance nurses' knowledge and skills. CNE for palliative care in Indonesian training programs has not been structurally established yet. It is fragmented in its application into some areas and has not been applied for the majority of areas in Indonesia.

Investigators aim to develop a palliative care training for PHC nurses using an online format. It will be done in several steps. Firstly, investigators are starting by conducting a review to collect information on what topics are suitable for PHC nurses. Secondly, investigators are developing modules and other educational tools (a virtual education package). Thirdly, those educational packages will be then evaluated by experts. Next, the education package will be integrated into eLOK (e-learning: open for knowledge sharing) at Universitas Gadjah Mada. After that, training for PHC nurses in Yogyakarta using eLOK will be conducted under the acronym: SPARK or Strengthening PAlliative caRe in the community by enhancing nurses' Knowledge (Sinau PAliatif Rame-rame karo eLOK). The effectiveness of SPARK will be measured with a Randomized Control Trial. Investigators will also collect more information on the feasibility of this program using qualitative data collection since investigators expect to refine this program to be applied in a larger area in Indonesia.

DETAILED DESCRIPTION:
Palliative care defines as an approach that improved the quality of life of patients and their family caregivers who are facing problems associated with life threatening (WHO, 2010). The definition is referring to any life-threatening illness such as cancer, dementia, heart failure, and so on. The number of people who needs palliative care is increasing significantly with the increasing number of older people and other degenerative diseases. In fact, more than 75%% people who died from serious health disease were in the developing countries (Spruyt, 2018; WHO, 2010).

In Indonesia, palliative care implementation has just started in 2007 under the ministry of health regulation: SK Menteri Kesehatan No 812/Menkes/SK/VII/2007 (Indonesia, 2007). According to this regulation, palliative care is recommended to be implemented in 5 provinces in Indonesia: Jakarta, Surabaya, Yogyakarta, Makasar dan Bali. It should be applied in all health care settings namely: hospital, primary care, and long term institution. However, the practical implementation in Indonesia has been slowly improved.

The first challenge is due to the insufficiently knowledge of palliative care of health care professionals. In Indonesia, palliative care has started in 2007, but it has just been integrated recently into health care curriculum. Another challenge is that palliative care team usually is formed in hospital based. Meanwhile, most patients who need palliative care are based at home. In the low middle income countries, like Indonesia, community plays an important role in palliative care. Therefore, health care professionals in the Primary Health Centre (PHC) need to be prepared for basic palliative care concept (Putranto, Mudjaddid, Shatri, Adli, & Martina, 2017).

In comparison to other countries in Asian regions, palliative care Indonesia is still slowly developed since Indonesia physician specialist in palliative care has not existed and the scarcity in the drugs regulation (Yamaguchi et al., 2014). Based on the worldwide report in 2015 by the Economist Intelligence Unit (EIU), amongst 80 countries, Indonesia ranked 53rd for palliative care implementation based several indicators: national policies, integration into health care services, hospice services and community engagement (Unit., 2015). Education and training for palliative care for Indonesian health care professional is lacking. Therefore, this should be conducted to accelerate the implementation of palliative care in Indonesia.

The investigators conducted previous study for palliative care implementation in PHC in Yogyakarta from 12 PHCs around Sleman, Kota Yogyakarta and Bantul. It showed that most nurses had not had enough information about palliative care. The concept of palliative care are mixed with other concept such as wound care, homecare and so forth (Unpublished, 2014). Although in Yogyakarta region, palliative care training for nurses and physicians have been performed regularly. However, these trainings were mostly included managerial staff and not the staff who are working directly with the patient. There is a limitation on transferring knowledge from those who attended trainings to those who directly contact with patients.

Conducting a training in a conventional way (face-to-face training) faces some challenges. Although it has plenty advantages as participants and trainee can spend some time to study, but the number of participants is limited due to time and budget. Also during this covid-19 pandemic situation, a conventional education session is hardly possible.

Knowing how important palliative care education for all health care professionals who work in the community, continuing nursing education is essential. In relation to the physical distancing regulation, an online learning can be the most possible solution in order to address this need. In this randomised control trial study, investigators attempt to test the effectiveness of an online learning program for palliative care for PHC nurses in Yogyakarta.

ELIGIBILITY:
Inclusion Criteria:

* - Nurses who currently work in Primary Health Center (PHC) in Yogyakarta, Indonesia, at least for one year;
* Able to access the Internet; and
* Willing to be part of the study.

Exclusion Criteria:

* Nurses working in PHC Yogyakarta but unable to provide consent due to some limitations (on leave, do not have enough time, do not have Internet access, temporary leaving job due to study commitment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
PHC nurse' knowledge | Week 0 (baseline), Week 5 (after intervention), Week 10 (follow up), Week 14 (follow up)
  Primary outcome of the current study is to measure the changes of the level of knowledge of PHC nurses. Investigators are using Palliative Care Quiz for Nursing Indonesian version (PCQN-i) from baseline to after intervention and to 4 and 8 weeks post intervention. This instrument (N=20 items) measures nurses' knowledge on palliative care which consists of 3 domains: philosophy and principles (4 items); pain and symptom management (13 items); and psychosocial and spiritual care (3 items). Items are responded to by 'true', 'false' and 'don't know' and each correct answer will score 1. The higher score will indicate the greater palliative care knowledge.

SECONDARY OUTCOMES:
PHC nurse's difficulty in palliative care | Week 0 (baseline), Week 5 (after intervention), Week 10 (follow up), Week 14 (follow up)
  Secondary aims are to measure the changes of perception of PHC nurses in the implementation of palliative care in the community using Palliative Care Difficulty Scale (PCDC). It is a validated tool to quantify the levels of difficulty when health professionals provide palliative care. This instrument (N=18 items) includes five subscales: expert support, alleviating symptoms, community coordination, communication in multidisciplinary teams and communication with patients and families. Each subscale has three items graded on a 5 point Likert-type scale from 1 = never to 5 = very much. A higher value means more perceived difficulties, with a possible score range from 1 to 5.
PHC nurse's practice report | Week 0 (baseline), Week 5 (after intervention), Week 10 (follow up), Week 14 (follow up)
  Another secondary aim is to measure the changes of reporting implementation of palliative care in the community using the Palliative Care Self-Reported Practice Scale. It is a validated tool to quantify the levels of adherence to recommended practices in palliative care (N=15 items). This scale is comprised of six sub scales graded on a 5 point Likert-type scale from never to very much. A higher value means closer adherence to recommended practices in palliative care, with possible score range from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Sinta Kristanti, PhD, Principal Investigator — Gadjah Mada University
Locations (1):
- Primary Health Center, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon the request to principle investigator
Supporting Information: Study Protocol
Time Frame: in 2022